CLINICAL TRIAL: NCT02817178
Title: Prospective Study for Validation of Immunological Biomarkers in Patients With Metastatic Colorectal Cancer
Brief Title: Study for Validation of Immunological Biomarkers in Patients With Metastatic Colorectal Cancer
Acronym: Epitopes-CRC02
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Epitopes-CRC02
Record Dates: First submitted 2016-06-27; First posted 2016-06-29 (Estimated); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

ARMS (1):
- Additional biological samples (Other): Additional blood samples will be realized specifically to the study at baseline, at 1 month, at 3 months, and 1 month after surgery (if applicable).
  Peripheral Blood Mononuclear Cell (PBMC) and plasma will be collected. Tissue tumor is collected during surgery if applicable.
  Interventions: Other: Additional biological samples

INTERVENTIONS:
Other: Additional biological samples — blood and tumor tissue samples

SUMMARY:
The investigators recently identified promiscuous HLA-DR-derived epitopes from the human telomerase reverse transcriptase (TERT) called universal cancer peptides (UCP), to study tumor-specific CD4+ T cell responses.

The investigators found high frequency of naturally occuring UCP-specific TH1 cells in long term survival of metastatic colorectal cancer (CRC) previously treated by 5 fluoro-uracil -oxaliplatin (Folfox) +/- bevacizumab regiment (Godet et al. OncoImmunology 2012 and unpublished data).

Epitopes-CRC02 is a French prospective multicenter study which will evaluate the post chemotherapy and post surgery modulation of host tumor-specific CD4 TH1 cell responses in metastatic colorectal cancer patients and their correlation with progression-free survival.

ELIGIBILITY:
Inclusion Criteria:

* Performance status ECOG-WHO 0, 1 or 2
* Metastatic colorectal cancer Histologically proved
* signed written informed consent

Exclusion Criteria:

* previous treatment (chemotherapy, targeted therapy, surgery) for metastatic disease
* history of autoimmune disease
* patients under immunotherapy systemic treatment or immunosuppressive drugs or stopped for less than 6 months to the enrollment in this study.
* corticoids ≥ 1mg/kg
* acute or chronic infectious disease during treatment or stopped for less than six months
* other malignancy within the last 5 years, except for adequately treated carcinoma in situ of the cervix or squamous carcinoma of the skin, or adequately controlled limited basal cell skin cancer.
* pregnancy, breast-feeding or absence of adequate contraception for fertile patients
* patient with any medical or psychiatric condition or disease which would make the patient inappropriate for entry into this study.
* patient under guardianship, curator or under the protection of justice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2017-06-11 (Actual); Study Completion 2020-07-06 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | date of first progression of the disease (within 3 years after the enrollment in the study)]
  time interval between the date of initiation of treatment and the date of first progression (local, remote [extent of the disease by RECIST v1.1] second cancer) or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Stefano KIM, Dr, Principal Investigator — CHU DE BESANCON
Locations (9):
- France (9):
  - Centre Hospitalier Régional Universitaire de Besançon, Besançon
  - Polyclinique de Franche-Comté, Besançon
  - Hôpitaux Civils de Colmar, Colmar
  - Centre Georges François Leclerc, Dijon
  - Hôpital Nord Franche-Comté, Montbéliard
  - Institut de Cancérologie de Lorraine, Nancy
  - Hôpital Européen Georges Pompidou, Paris
  - Centre Paul Strauss, Strasbourg
  - Centre Hospitalier Universitaire de Tours, Tours

REFERENCES:
- [Derived] Kroemer M, Turco C, Spehner L, Viot J, Idirene I, Bouard A, Renaude E, Deschamps M, Godet Y, Adotevi O, Limat S, Heyd B, Jary M, Loyon R, Borg C. Investigation of the prognostic value of CD4 T cell subsets expanded from tumor-infiltrating lymphocytes of colorectal cancer liver metastases. J Immunother Cancer. 2020 Nov;8(2):e001478. doi: 10.1136/jitc-2020-001478. PMID 33229508